CLINICAL TRIAL: NCT01706432
Title: Biologic Endpoints in the Annihilation of Metastases for Oligometastasis (BEAM ON)
Brief Title: Hypofractionated Image Guided Radiation Therapy in Treating Patients With Stage IV Breast Cancer
Status: Completed | Type: Observational
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: 16802B; NCI-2011-03193 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-10-05; First posted 2012-10-15 (Estimated); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Central Nervous System Metastases; Invasive Ductal Breast Carcinoma; Invasive Ductal Breast Carcinoma With Predominant Intraductal Component; Invasive Lobular Breast Carcinoma; Invasive Lobular Breast Carcinoma With Predominant in Situ Component; Liver Metastases; Lobular Breast Carcinoma in Situ; Lung Metastases; Male Breast Cancer; Medullary Ductal Breast Carcinoma With Lymphocytic Infiltrate; Mucinous Ductal Breast Carcinoma; Papillary Ductal Breast Carcinoma; Recurrent Breast Cancer; Stage IV Breast Cancer; Tubular Ductal Breast Carcinoma; Tumors Metastatic to Brain
MeSH Terms: conditions — Carcinoma, Ductal, Breast; Carcinoma, Lobular; Breast Carcinoma In Situ; Breast Neoplasms, Male; Breast Neoplasms; Brain Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All participants: Patients will undergo standard of care radiation therapy and have research blood samples collected at following time points:
  * pre-treatment
  * 3-4 weeks post-treatment
  * every 9-12 weeks post-treatment for 1 year
  Interventions: Radiation: hyperfractionated radiation therapy; Other: laboratory biomarker analysis; Radiation: stereotactic radiosurgery

INTERVENTIONS:
Radiation: hyperfractionated radiation therapy — Undergo hypofractionated radiation therapy
Other: laboratory biomarker analysis — Correlative studies
Radiation: stereotactic radiosurgery — Undergo stereotactic radiosurgery

SUMMARY:
This pilot clinical trial studies new ways to monitor the impact of hypofractionated image guided radiation therapy in treating patients with stage IV breast cancer. Radiation therapy uses high energy x rays to kill tumor cells. Giving radiation therapy in different ways may kill more tumor cells.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven diagnosis of breast cancer (invasive ductal, lobular, medullary, papillary, colloid, tubular)
* Completion of standard of care treatment for local and regional disease with no known residual
* American Joint Committee on Cancer (AJCC) (6th edition, 2002) Stage IV ( Any T, Any N, M1) based upon the following minimum diagnostic workup:
* History/physical examination within 8 weeks prior to registration
* Computed tomography (CT), magnetic resonance imaging (MRI) and/or positron emission tomography (PET) CT of the whole body within 60 days prior to registration
* MRI of the brain, if clinically indicated
* Documentation of 1-5 sites of metastatic tumor; each individual site of tumor must be =< 10 cm or < 500 cc volume and amenable to radiation therapy as seen on standard imaging (CT, MRI, bone scan)
* Pathology from at least one metastatic site confirming breast primary is recommended
* Zubrod performance status =< 2 (Karnofsky >= 60%)
* Absolute neutrophil count (ANC) >= 1,800 cells/mm^3
* Platelets >= 100,000 cells/mm^3
* Hemoglobin >= 8.0 g/dl (Note: The use of transfusion or other intervention to achieve hemoglobin [Hgb] >= 8.0 g/dl is acceptable)
* Total bilirubin within institutional limits
* Albumin > 2.9 g/dl
* Alkaline phosphatase < 2.5x upper limit of normal (ULN)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 2.5 x ULN
* Room air saturation (saturated oxygen [Sa02]) > 90%
* Life expectancy > 3 months
* Patient complete study specific informed consent process and sign consent form prior to study entry
* Patients with prior metastatic treatment are eligible if they have been disease free for > 3 years; participants may receive hormonal and Herceptin treatment at any time

Exclusion Criteria:

* Patients are ineligible if they have had prior treatment for their metastatic disease within 3 years
* Prior radiotherapy that would result in overlap of radiation therapy fields
* Co-existing or prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 3 years (for example, carcinoma in situ of the breast, oral cavity, or cervix are all permissible)
* Severe, active co-morbidity, defined as follows:
* Clinically significant pulmonary dysfunction, cardiomyopathy, any history of clinically significant congestive heart failure (CHF), unstable angina pectoris, or cardiac arrhythmia
* Transmural myocardial infarction within the last 6 months
* Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration
* Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of registration
* Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects; note, however, that laboratory tests for liver function and coagulation parameters are not required for entry into this protocol
* Acquired Immune Deficiency Syndrome (AIDS) based upon current Centers for Disease Control (CDC) definition; note, however, that human immunodeficiency virus (HIV) testing is not required for entry into this protocol; the need to exclude patients with AIDS from this protocol is necessary because the treatments involved in this protocol may be significantly immunosuppressive; protocol-specific requirements may also exclude immunocompromised patients
* Pregnancy, breast feeding or women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception during treatment and for at least three months following completion; this exclusion is necessary because the treatment involved in this study may be significantly teratogenic
* Prior treatment with anti-angiogenic therapy
* Significant atelectasis such that CT definition of the gross tumor volume (GTV) is difficult to determine
* Exudative, bloody or cytologically malignant effusions
* Evidence of pleural or pericardial effusion prior to study start; patients with pleural effusion that is transudative, cytologically negative, and non-bloody are eligible; if a pleural effusion is too small for diagnostic thoracentesis, the patient will be eligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving radiation treatment for breast cancer.
Sampling Method: Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2009-06-15 (Actual); Primary Completion 2024-01-22 (Actual); Study Completion 2024-01-22 (Actual)

PRIMARY OUTCOMES:
Change in the number of circulating tumor cells | At baseline, 3-4 weeks post-treatment, and every 9-12 weeks for one year

SECONDARY OUTCOMES:
Progression free survival | 5 years
Overall survival | 5 years
Side effects of hypofractionated image guided radiotherapy | During treatment (about 21 days)
Number of patients with IRDS in tumor sample | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Steven Chmura, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, North Chicago, Illinois, United States